CLINICAL TRIAL: NCT03984409
Title: A Dietary Source of Potassium Citrate to Resolve Hypocitraturia and Aciduria in Patients With a History of Nephrolithiasis
Brief Title: A Dietary Source of Potassium Citrate to Resolve Hypocitraturia and Aciduria in Patients With Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Large, Principal Investigator, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1903221743
Record Dates: First submitted 2019-05-22; First posted 2019-06-13 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Potassium Citrate

STUDY DESIGN:
Intervention Model Description: Group 1 kcit x 7 days ↓ Litholink on day 7
  ↓ off therapy x 7 days
  ↓ OJ 500 ML + 1.5L water /day x 7 days
  ↓ Litholink on day 7
  ↓ OJ 1000 ML + 1L water /day x 7 days
  ↓ Litholink on day 7 Return to kcit therapy
  Group 2 OJ 500 ML + 1.5L water /day x 7 days ↓ Litholink on day 7
  ↓ OJ 1000 ML + 1L water /day x 7 days
  ↓ Litholink on day 7
  ↓ off therapy x 7 days
  ↓ kcit x 7 days
  ↓ Litholink on day 7 Continue on kcit therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Potassium citrate x 7days Off therapy x 7 days 500 mL low calorie orange juice beverage x 7 days 1000 mL low calorie orange juice beverage x 7 days Return to potassium citrate therapy Litholink urine collection to be performed after each 7 days treatment
  Interventions: Dietary Supplement: Kroger low calorie orange juice beverage
- Group 2 (Active Comparator): 500 mL low calorie orange juice beverage x 7 days 1000 mL low calorie orange juice beverage x 7 days Off therapy x 7 days Potassium citrate x 7days Continue on potassium citrate therapy Litholink urine collection to be performed after each 7 days treatment
  Interventions: Dietary Supplement: Kroger low calorie orange juice beverage

INTERVENTIONS:
Dietary Supplement: Kroger low calorie orange juice beverage — Kroger low calorie orange juice beverage will be consumed for 7 days followed by a 24 hour urine collection with Litholink to see if urine alkalization similar to potassium citrate can be achieved
  Other Names: potassium citrate

SUMMARY:
Patients with nephrolithiasis and evidence of hypocitraturia or aciduria who would otherwise be started on potassium citrate, can achieve similar urine alkalization with 500-1000 mL of daily low calorie orange juice consumption.

DETAILED DESCRIPTION:
Potassium Citrate (kcit) has long been utilized by physicians to combat stone formation in patients with hypocitraturia or aciduria. The most common obstacle to patient compliance with this medication has historically been dosing frequency, pill size, dyspepsia, and its familiar unpleasant taste. However, rampant increases in drug pricing by pharmaceutical companies, that have achieved market control of the drug supply, are triggering non-compliance in the subset of stone patients who depend on potassium citrate therapy to prevent stone recurrence.

Previous research has shown that certain commercially available beverages contain alkali citrate, of which orange juice (OJ) has the highest reported concentrations of potassium citrate based on ion chromatography. Unfortunately, the high sugar content of orange juice excludes its potential use as a dietary alternative to prescription potassium citrate. Recently, major beverage companies (Pepsi, Coca Cola) have release low calorie beverages with equivalent citrate content but with 50% less sugar. In early 2018 the investigaotrs performed ion-chromatography on various consumer beverages and validated that low calorie orange juice provided equivalent alkali citrate and malate to standard orange juice. The ion-chromatography also showed that the total amount of alkali/liter was greater in low calorie orange juice compared to crystal light lemon flavored. Currently, crystal light lemon is recommended as the next best option to water for recurrent stone formers with low urine volume production and hypocitraturia or aciduria (https://kidneystones.uchicago.edu/price-of-potassium-citrate/). However, there is a concern that the citrate within lemon based beverages is predominantly in an acidic form and thus has less potential to provide clinically affective levels of alkali despite a favorable alkali profile on ion chromatography.

Since low calorie orange juice was identified as a potential sources for citrate and alkali, the investigators wanted to show that consumption of the beverages resulted in desirable changes in urinary pH and citrate levels without negatively affecting patient well-being. Ten (10) volunteers drank standardized quantities of water, crystal light lemon juice, and two low calorie orange juices. After 7 days of beverage consumption the participants performed a 24 hour urine collection which was performed by an independent laboratory. The participants also maintained a diary of dietary (both food and drink) intake in addition to the trial beverages. The data from the study is very promising with desired changes in urinary pH and citrate levels with consumption of the low calorie orange juice. Minimal side effects were noted from consuming the low calorie orange juice except with Tropicana50 based on journals. It was determined that the artificial sweetener in TRP50 was the causative agent for GI symptoms and headaches. The preferred brand based on volunteer diaries was a generic brand by Kroger® low calorie orange beverage.

Our data suggests that low calorie orange juice has the potential to improve compliance rates with alkali therapy amongst recurrent stone formers. Stone prevention is key to reducing long-term sequelae of repeat surgical intervention such as iatrogenic genitourinary strictures, infections, and end organ damage. Additionally, there is a large cost savings potential with stone prevention by reducing hospital stays, surgical procedures, and missed work days due to stone disease. While daily low calorie orange juice may not completely supplant prescription potassium citrate therapy, it may be a favorable adjunct to reduce cost associated with potassium citrate and increase compliance rates by reducing the dose required to clinically relevant alkalization of the urine. Our hypothesis, is that patients with nephrolithiasis and evidence of hypocitraturia or aciduria who would otherwise be started on potassium citrate, can achieve similar urine alkalization with 500-1000 mL of daily low calorie orange juice consumption.

ELIGIBILITY:
Inclusion Criteria:

* • Between 18 and 75 year of age.

  * History of kidney stone disease with available stone analysis
  * Evidence of aciduria or hypocitraturia on 24 hour urinalysis (24 hr citrate male <450 mg/day female <550 mg/day) or aciduria (urine pH < 5.8)
  * Ability to drink Kroger low calorie orange juice beverage
  * If subject with history of diabetes mellitus, must have HgA1c < 7.5 and willing to check daily blood sugars.

Exclusion Criteria:

* • Less than 18 or older than 75 years of age

  * Allergies to low calorie orange juice, including intolerance because of side effects including (but not limited to): gastrointestinal symptoms, headaches, weight gain, unable to drink because of taste.
  * Poorly controlled diabetic (HgA1c >7.5)
  * No evidence of hypocitraturia or aciduria on 24 hour urinalysis
  * Unable to afford potassium citrate therapy or tolerate medication because of side effects.
  * Unwilling to perform 3 24-hour urine collections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Urine alkalization from Kroger low calorie orange juice beverage | 9 weeks from enrollment
  The primary endpoint of interest will be the changes in urinary citrate while consuming Kroger low calorie orange juice beverage compared to potassium citrate therapy.
Urine alkalization from Kroger low calorie orange juice beverage | 9 weeks from enrollment
  The primary endpoint of interest will be the changes in urinary pH while consuming Kroger low calorie orange juice beverage compared to potassium citrate therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Large, MD, Principal Investigator — Indiana University Health
Locations (2):
- United States (2):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Health Physicians Urology, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No